CLINICAL TRIAL: NCT02797522
Title: A Sequential Phase 1a/1b Dose-Escalating Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of ARC-521 in Normal Adult Volunteers and Patients With Chronic Hepatitis B
Brief Title: A Study of ARC-521 Injection in Normal Adult Volunteers and Patients With Chronic Hepatitis B (CHB)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision to discontinue trial
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARC5211001
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Histamine Antagonists; Acetaminophen; entecavir; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (11):
- NHV Participants: Cohort 1 (Experimental): NHV participants administered a single dose of ARC-521 Injection at a dose of 0.6 mg/kg.
  Interventions: Drug: ARC-521 Injection; Drug: antihistamine; Drug: acetaminophen
- NHV Participants: Cohort 2 (Experimental): NHV participants administered a single dose of ARC-521 Injection at a dose of 1 mg/kg.
  Interventions: Drug: ARC-521 Injection; Drug: antihistamine; Drug: acetaminophen
- NHV Participants: Cohort 3 (Experimental): NHV participants administered a single dose of ARC-521 Injection at a dose of 2 mg/kg.
  Interventions: Drug: ARC-521 Injection; Drug: antihistamine; Drug: acetaminophen
- NHV Participants: Cohort 4 (Experimental): NHV participants administered a single dose of ARC-521 Injection at a dose of 4 mg/kg.
  Interventions: Drug: ARC-521 Injection; Drug: antihistamine; Drug: acetaminophen
- NHV Participants: Cohort 5 (Experimental): NHV participants administered a single dose of ARC-521 Injection at a dose of 5 mg/kg.
  Interventions: Drug: ARC-521 Injection; Drug: antihistamine; Drug: acetaminophen
- NHV Participants: Cohort 6 (Experimental): NHV participants administered a single dose of ARC-521 Injection at a dose of 6 mg/kg.
  Interventions: Drug: ARC-521 Injection; Drug: antihistamine; Drug: acetaminophen
- NHV Participants: Placebo (Placebo Comparator): NHV participants administered 0.9% normal saline to match ARC-521 Injection at doses of 0.6, 1, 2, 4, 5 and 6 mg/kg.
  Interventions: Other: Placebo; Drug: antihistamine; Drug: acetaminophen
- CHB Participants: Cohort 3b (Experimental): Treatment-naive participants with CHB administered 3 doses of ARC-521 Injection at 2 mg/kg once every 4 weeks. Participants are treatment-naive if they have not been on continual nucleoside analog (NUC) therapy (any NUC) for at least 6 months prior to screening (or have never been on NUCs).
  Interventions: Drug: ARC-521 Injection; Drug: antihistamine; Drug: acetaminophen
- CHB Participants: Cohort 4b (Experimental): Treatment-naive participants with CHB administered 3 doses of ARC-521 Injection at 4 mg/kg once every 4 weeks. Participants are treatment-naive if they have not been on continual NUC therapy (any NUC) for at least 6 months prior to screening (or have never been on NUCs).
  Interventions: Drug: ARC-521 Injection; Drug: antihistamine; Drug: acetaminophen
- CHB Participants: Cohort 3c (Experimental): Participants with CHB currently on NUCs (entecavir or tenofovir for at least 6 months) administered 3 doses of ARC-521 Injection at 2 mg/kg once every 4 weeks.
  Interventions: Drug: ARC-521 Injection; Drug: antihistamine; Drug: acetaminophen; Drug: entecavir; Drug: tenofovir
- CHB Participants: Cohort 4c (Experimental): Participants with CHB currently on NUCs (entecavir or tenofovir for at least 6 months) administered 3 doses of ARC-521 Injection at 4 mg/kg once every 4 weeks.
  Interventions: Drug: ARC-521 Injection; Drug: antihistamine; Drug: acetaminophen; Drug: entecavir; Drug: tenofovir

INTERVENTIONS:
Drug: ARC-521 Injection
  Arms: CHB Participants: Cohort 3b; CHB Participants: Cohort 3c; CHB Participants: Cohort 4b; CHB Participants: Cohort 4c; NHV Participants: Cohort 1; NHV Participants: Cohort 2; NHV Participants: Cohort 3; NHV Participants: Cohort 4; NHV Participants: Cohort 5; NHV Participants: Cohort 6
Other: Placebo — 0.9% normal saline
  Arms: NHV Participants: Placebo
Drug: antihistamine — Approximately two hours prior to ARC-521 or placebo administration, participants will be pre-treated with an oral antihistamine, selected by the investigator from the list of approved antihistamines that is available in that country. Approved antihistamines are: diphenhydramine 50 mg by mouth (PO), chlorpheniramine 8 mg PO, or hydroxyzine 50 mg PO.
Drug: acetaminophen — Approximately two hours prior to ARC-521 or placebo administration, participants will be pre-treated with acetaminophen (500 - 1000 mg PO, per local strength availability).
Drug: entecavir — Participants take entecavir OR tenofovir daily throughout the study.
  Arms: CHB Participants: Cohort 3c; CHB Participants: Cohort 4c
Drug: tenofovir — Participants take entecavir OR tenofovir daily throughout the study.
  Arms: CHB Participants: Cohort 3c; CHB Participants: Cohort 4c

SUMMARY:
Normal healthy volunteer (NHV) participants will enroll sequentially into a total of 6 escalating dose levels (6 subjects per dose level), randomized to receive a single dose of ARC-521 Injection or placebo. The maximum study duration for NHVs is approximately 21 weeks.

Hepatitis B e Antigen (HBeAg)-negative participants with (CHB) will enroll sequentially into 3 dose levels (8 patients per dose level) to receive multiple doses of open label ARC-521 Injection. For each CHB participant the maximum study duration is approximately 37 weeks.

DETAILED DESCRIPTION:
Phase 1a/1b multicenter dose-escalation study of ARC-521 Injection in normal healthy volunteers and patients with CHB. Eligible participants who have signed an Ethics Committee (EC)/Institutional Review Board (IRB) approved informed consent form and have met all of the protocol eligibility criteria.

Patients will undergo the following evaluations at regular intervals during the study: medical history, physical examinations, vital sign measurements (blood pressure, heart rate, respiratory rate, and temperature), weight, adverse events assessment (AEs), concomitant medications/therapies assessment, electrocardiograms (ECGs), telemetry [NHVs only], measures of hepatic fibrosis [CHBs only], blood sample collection for hematology, coagulation, chemistry, Pharmacokinetics (PK) [NHVs only], metabolic analysis [NHVs only], exploratory Pharmacodynamic (PD) measures, urinalysis, hepatitis B virus (HBV) serology, immunogenicity, Follicle Stimulating Hormone (FSH) testing (post-menopausal females) and pregnancy testing for females of childbearing potential. Clinically significant changes including AEs will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the patient is lost to follow-up. Prior to enrollment there is a 60 day screening period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 55 years of age inclusive (NHVs) or 18-65 years of age inclusive (CHBs), at the time of informed consent
* Able to provide written informed consent prior to the performance of any study specific procedures
* Body mass index (BMI) between 19.0 and 35.0 kg/m2, inclusive
* A 12-lead ECG at Screening and pre-dose assessment that, in the opinion of the investigator, has no abnormalities that compromise participant's safety in this study
* Must use 2 effective methods of contraception (double barrier contraception or hormonal contraceptive along with a barrier contraceptive (both male and female partners)
* Have suitable venous access for blood sampling
* No abnormal finding of clinical relevance at the Screening evaluation (NHVs only)
* Have a diagnosis of HbeAg-negative chronic HBV infection (CHB patients only)
* Treatment-naive or currently on entecavir/tenofovir for 6 months or longer

Exclusion Criteria:

* Pregnant or lactating
* Acute signs of hepatitis/other infection at Screening or at baseline
* Use within last 14 days or anticipated requirement for anticoagulants, systemic corticosteroids, immunomodulators, or immunosuppressants
* Use of prescription medication within 14 days prior to study treatment that in the opinion of the PI or the Sponsor would interfere with study conduct.
* Known diagnosis of non-alcoholic steatohepatitis [NHVs only] or familial hypercholesterolemia
* Taking interferon alpha (INFalpha) within 6 months of screening [CHBs only]
* History of poorly controlled autoimmune disease or history of autoimmune hepatitis
* Human immunodeficiency virus (HIV) infection
* Seropositive for HBV (NHVs only) or hepatitis C virus (HCV), and/or history of delta virus hepatitis
* Hypertension defined as blood pressure > 170/100 mmHg at screening [NHVs only]
* A history of cardiac rhythm disturbances
* Family history of congenital long QT syndrome, Brugada syndrome or unexplained sudden cardiac death
* Symptomatic heart failure, unstable angina, myocardial infarction, severe cardiovascular disease within 6 months prior to study entry
* History of malignancy within the last 5 years except for adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer
* History of major surgery within 3 months of Screening
* Regular use of alcohol within one month prior to the Screening visit (more than fourteen units of alcohol per week)
* Evidence of severe systemic acute inflammation, sepsis, or hemolysis [NHVs only]
* Use within 3 months of illicit drugs (cocaine, phencyclidine [PCP], 3,4-methylenedioxymethamphetamine [MDMA], others) or positive test for drugs of abuse at screening.
* History of allergy to bee venom or history of severe hypersensitivity reaction, such as anaphylaxis
* Use of an investigational agent or device within 30 days prior to dosing or current participation in an investigational study
* Clinically significant history of any alcoholic liver disease, cirrhosis, Wilson's disease, hemochromatosis, or alpha-1 antitrypsin deficiency, liver or kidney disease
* Clinically significant history/presence of poorly controlled or decompensated neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, metabolic, or other uncontrolled systemic disease
* Blood donation (500 mL) within 7 days prior to study treatment administration [NHVs only]
* History of fever (>38.0ºC/100.4ºF) within 2 weeks of Screening [NHVs only]
* Any concomitant medical or psychiatric condition or social situation that impacts compliance or involves additional safety risk
* History of coagulopathy (including deep vein thrombosis and pulmonary embolism) or stroke within 6 months of baseline, and/or concurrent anticoagulant medication(s)
* Presence of cholangitis, cholecystitis, cholestasis, or duct obstruction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site 1, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NHV Participants: Cohort 1: Normal healthy volunteer (NHV) participants administered a single dose of ARC-521 Injection at a dose of 0.6 mg/kg.
- CHB Participants: Cohort 3b: Treatment-naive participants with chronic hepatitis B (CHB) administered 3 doses of ARC-521 Injection at 2 mg/kg once every 4 weeks. Participants are treatment-naive if they have not been on continual nucleoside analog (NUC) therapy (any NUC) for at least 6 months prior to screening (or have never been on NUCs).
Period: Overall Study
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo | CHB Participants: Cohort 3b | CHB Participants: Cohort 4b | CHB Participants: Cohort 3c | CHB Participants: Cohort 4c
Started | 4 | 4 | 4 | 4 | 4 | 4 | 12 | 4 | 2 | 4 | 1
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 12 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 4 | 1
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- CHB Participants: Cohort 3b: Treatment-naive participants with CHB administered 3 doses of ARC-521 Injection at 2 mg/kg once every 4 weeks. Participants are treatment-naive if they have not been on continual NUC therapy (any NUC) for at least 6 months prior to screening (or have never been on NUCs).
- CHB Participants: Cohort 4b: Treatment-naive participants with CHB administered 3 doses of ARC-521Injection at 4 mg/kg once every 4 weeks. Participants are treatment-naive if they have not been on continual NUC therapy (any NUC) for at least 6 months prior to screening (or have never been on NUCs).
- Total: Total of all reporting groups
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo | CHB Participants: Cohort 3b | CHB Participants: Cohort 4b | CHB Participants: Cohort 3c | CHB Participants: Cohort 4c | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 12 | 4 | 2 | 4 | 1 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (8.26) | 27.8 (10.90) | 23.3 (3.30) | 22.5 (1.29) | 22.3 (3.59) | 23.5 (4.04) | 28.3 (5.69) | 46.3 (10.63) | 44.5 (14.85) | 44.3 (3.69) | 36.0 (NA) — 1 participant in cohort | 30.0 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 1 | 1 | 3 | 7 | 0 | 0 | 0 | 1 | 18
  Male | 3 | 1 | 3 | 3 | 3 | 1 | 5 | 4 | 2 | 4 | 0 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs): Healthy Volunteers
Description: An adverse event (AE) is any untoward medical occurrence which does not necessarily have a causal relationship with this treatment. A serious AE is any AE that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is a medically important event or reaction.Events were categorized as mild, moderate or severe. TEAEs were defined as all AEs starting or worsening after commencement of treatment with investigational product. A treatment-related TEAE was one whose relationship to treatment was noted as unlikely, possibly, or probably related.
Time Frame: From first dose of study drug through Day 29 (± 1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 12
Participants
  >/= 1 TEAE | 1 | 2 | 3 | 4 | 3 | 2 | 10
  >/= 1 Serious TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >/= 1 Related TEAE | 0 | 0 | 1 | 2 | 2 | 1 | 3
  >/= 1 Related Serious TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With TEAEs: CHB Participants
Description: An AE is any untoward medical occurrence which does not necessarily have a causal relationship with this treatment. A serious AE is any AE that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is a medically important event or reaction.Events were categorized as mild, moderate or severe. TEAEs were defined as all AEs starting or worsening after commencement of treatment with investigational product. A treatment-related TEAE was one whose relationship to treatment was noted as unlikely, possibly, or probably related.
Time Frame: From first dose of study drug through Day 142 (± 3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | CHB Participants: Cohort 3b | CHB Participants: Cohort 4b | CHB Participants: Cohort 3c | CHB Participants: Cohort 4c
Number analyzed (Participants) | 4 | 2 | 4 | 1
Participants
  >/= 1 TEAE | 2 | 1 | 4 | 1
  >/= 1 Serious TEAE | 0 | 1 | 0 | 0
  >/= 1 Related TEAE | 0 | 1 | 2 | 0
  >/= 1 Related Serious TEAE | 0 | 1 | 0 | 0

3. Primary Outcome: Pharmacokinetics of ARC-521 Injection: Area Under the Plasma-Concentration-Time Curve From Time 0-24 Hours (AUC0-24), Healthy Volunteers
Time Frame: Through 48 hours post-dose on Day 1
Population: Analysis was not planned or conducted per statistical analysis plan (SAP) due to study termination.
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Pharmacokinetics of ARC-521 Injection: Area Under the Plasma-Concentration-Time Curve From Time 0 to the Last Quantifiable Plasma Concentration (AUClast), Healthy Volunteers
Time Frame: Through 48 hours post-dose on Day 1
Population: Analysis was not planned or conducted per SAP due to study termination.
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Pharmacokinetics of ARC-521 Injection: Area Under the Plasma-Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUCinf), Healthy Volunteers
Time Frame: Through 48 hours post-dose on Day 1
Population: Analysis was not planned or conducted per SAP due to study termination.
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Pharmacokinetics of ARC-521 Injection: Maximum Observed Plasma Concentration (Cmax), Healthy Volunteers
Time Frame: Through 48 hours post-dose on Day 1
Population: Analysis was not planned or conducted per SAP due to study termination.
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Pharmacokinetics of ARC-521 Injection: Clearance (CL), Healthy Volunteers
Time Frame: Through 48 hrs post-dose on Day 1
Population: Analysis was not planned or conducted per SAP due to study termination.
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Pharmacokinetics of ARC-521 Injection: Apparent Volume of Distribution (V), Healthy Volunteers
Time Frame: Through 48 hours post-dose on Day 1
Population: Analysis was not planned or conducted per SAP due to study termination.
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Pharmacokinetics of ARC-521 Injection: Terminal Elimination Rate Constant (Kel), Healthy Volunteers
Time Frame: Through 48 hours post-dose on Day 1
Population: Analysis was not planned or conducted per SAP due to study termination.
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Pharmacokinetics of ARC-521 Injection: Terminal Elimination Half-Life (t1/2), Healthy Volunteers
Time Frame: Through 48 hours post-dose on Day 1
Population: Analysis was not planned or conducted per SAP due to study termination.
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

11. Primary Outcome: Change Over Time in Viral Antigens and DNA in CHB Participants as a Measure of Activity of ARC-521 Injection
Time Frame: Baseline to Day 142
Population: Analysis was not planned or conducted per SAP due to study termination.
Arm/Group | CHB Participants: Cohort 3b | CHB Participants: Cohort 4b | CHB Participants: Cohort 3c | CHB Participants: Cohort 4c
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Change Over Time in Cytokine Levels After Single and Multiple Doses of ARC-521 Injection
Time Frame: Through 24 hours post-dose (Day 1 for NHVs, and Days 1, 29 & 57 for CHB participants)
Population: Analysis was not planned or conducted per SAP due to study termination.
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo | CHB Participants: Cohort 3b | CHB Participants: Cohort 4b | CHB Participants: Cohort 3c | CHB Participants: Cohort 4c
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Change Over Time in Complement Levels After Single and Multiple Doses of ARC-521 Injection
Time Frame: Through 24 hours post-dose (Day 1 for NHVs, and Days 1, 29 & 57 for CHB participants)
Population: Analysis was not planned or conducted per SAP due to study termination.
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo | CHB Participants: Cohort 3b | CHB Participants: Cohort 4b | CHB Participants: Cohort 3c | CHB Participants: Cohort 4c
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: NHV: from first dose of study drug through Day 29 (± 1 days); CHB participants:from first dose of study drug through Day 142 (± 3 days)
Arm/Group | NHV Participants: Cohort 1 | NHV Participants: Cohort 2 | NHV Participants: Cohort 3 | NHV Participants: Cohort 4 | NHV Participants: Cohort 5 | NHV Participants: Cohort 6 | NHV Participants: Placebo | CHB Participants: Cohort 3b | CHB Participants: Cohort 4b | CHB Participants: Cohort 3c | CHB Participants: Cohort 4c
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/12 | 0/4 | 1/2 | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 1/4 | 2/4 | 3/4 | 4/4 | 3/4 | 2/4 | 10/12 | 2/4 | 0/2 | 4/4 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NHV Participants: Cohort 1 (N=4) | NHV Participants: Cohort 2 (N=4) | NHV Participants: Cohort 3 (N=4) | NHV Participants: Cohort 4 (N=4) | NHV Participants: Cohort 5 (N=4) | NHV Participants: Cohort 6 (N=4) | NHV Participants: Placebo (N=12) | CHB Participants: Cohort 3b (N=4) | CHB Participants: Cohort 4b (N=2) | CHB Participants: Cohort 3c (N=4) | CHB Participants: Cohort 4c (N=1)
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NHV Participants: Cohort 1 (N=4) | NHV Participants: Cohort 2 (N=4) | NHV Participants: Cohort 3 (N=4) | NHV Participants: Cohort 4 (N=4) | NHV Participants: Cohort 5 (N=4) | NHV Participants: Cohort 6 (N=4) | NHV Participants: Placebo (N=12) | CHB Participants: Cohort 3b (N=4) | CHB Participants: Cohort 4b (N=2) | CHB Participants: Cohort 3c (N=4) | CHB Participants: Cohort 4c (N=1)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Ear deformity acquired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The ARC-521 Injection development program was terminated early for regulatory and business reasons secondary to findings occurring in a non-clinical toxicology study. Program termination was not due to safety findings in humans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No